CLINICAL TRIAL: NCT06759272
Title: Pharmacogenomic Markers of Clopidogrel Resistance in Malaysian CAD Patients: Clinical Efficacy and Economic Evaluation of CYP2C19 Genotype-Guided Therapy
Brief Title: Impact of CYP2C19 Genotype-guided Approach in Antiplatelet Therapy on Platelet Reactivity Index Among Coronary Artery Disease (CAD) Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nur Hafizah Annezah binti Utuh (Other)
Responsible Party: Sponsor-Investigator, Nur Hafizah Annezah binti Utuh, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 311224
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arterial Disease (CAD); ACS (Acute Coronary Syndrome); SCAD
Keywords: CYP2C19 genotype-guided antiplatelet therapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Precision Medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intervention group (Experimental): Pre-emptive genetic testing will be done on the patients allocated randomly to the intervention group after obtaining their consent. The clinical decision making on the antiplatelet (either clopidogrel or ticagrelor) will be done based on the presence of genetic markers CYP2C19*2 and CYP2C19*3, according to the latest Clinical Pharmacogenetics Implementation Consortium (CPIC) 2022 guideline. Patients who are identified to have reduced function CYP2C19 allele will receive 90 mg ticagrelor and patients with wild-type CYP2C19 allele will receive clopidogrel 75 mg in the next scheduled dose.
  Interventions: Genetic: CYP2C19 genotype-guided antiplatelet therapy
- Universal Clopidogrel (No Intervention): All patients in the control group 1 will receive clopidogrel (300 mg loading dose to 75 mg daily maintenance dose) without any genetic screening done for 30 days.
- Universal Ticagrelor (No Intervention): All patients in the control group 2 will ticagrelor (180 mg loading dose to 90 mg twice daily as maintenance dose) without any genetic screening done for 30 days.

INTERVENTIONS:
Genetic: CYP2C19 genotype-guided antiplatelet therapy — A panel of genes including CYP2C19*2 (rs4244285) and CYP2C19*3 (rs4986893) will be genotyped using the real-time PCR and the expected turnover time will be 48 hours. Patients who are identified to have reduced function CYP2C19 allele will receive 90 mg ticagrelor and patients with wild-type CYP2C19 allele will receive clopidogrel 75 mg in the next scheduled dose. The switching done from clopidogrel to ticagrelor is supported by Antiplatelet Therapy Switching Clinician Guideline, whereby in the maintenance or low risk phase, there is generally no need to administer a loading dose of ticagrelor; one can switch directly to ticagrelor maintenance dose 24 hours after the last dose of clopidogrel
  Other Names: CYP2C19 screening test; Precision medicine
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if the pilot intervention of CYP2C19 genotype-guided antiplatelet therapy works to reduce the occurrence of cardiovascular events after Percutaneous Coronary Intervention (PCI) done in coronary artery disease patients. It will also learn about the comparison between clopidogrel and ticagrelor.

The main questions it aims to answer are:

To compare the impact of CYP2C19 genotype-guided antiplatelet therapy, universal use of clopidogrel and ticagrelor treatment on platelet reactivity.

To compare the impact of CYP2C19 genotype-guided antiplatelet therapy, universal use of clopidogrel and ticagrelor treatment on the risk of major adverse cardiovascular events (MACE) among newly recruited stable CAD patients.

Participants will:

Take drug clopidogrel or ticagrelor, based on the random group allocation every day for 1 month. One group of patients will undergone CYP2C19 genetic test for genotype-guided antiplatelet therapy, whether clopidogrel or ticagrelor.

Visit the clinic post 30 days of PCI for follow-ups and platelet function tests.

DETAILED DESCRIPTION:
Clopidogrel, a prodrug that inhibits platelet aggregation, is widely used in patients undergoing percutaneous coronary interventions to prevent recurrent cardiovascular events. However, clopidogrel resistance has emerged as a great concern, whereby it causes inadequate platelet inhibition and leads to antiplatelet treatment failure with prevalence as high as 44% in Asian population. Due to various established evidence from pharmacogenomics studies, US FDA has issued a black-box warning notifying that CYP2C19 polymorphisms may impaired the ability of a patient to convert clopidogrel into its active metabolite. Currently, the availability of newer P2Y12 receptor inhibitors has prompted medical professionals to consider genotype-guided treatment, which may include escalation or de-escalation of the antiplatelet based on CYP2C19 genetic result. We hypothesize that CYP2C19 genotype guided therapy will reduce the occurrence of MACE and improve platelet reactivity to prevent clopidogrel resistance. The estimated sample size required for pilot intervention study is 120 patients. Knowledge of potential pharmacogenetic markers for clopidogrel resistance, clinical efficacy and cost evaluation of genotype-guided antiplatelet therapy will provide a comprehensive insight into adopting such approach in a real routine clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Aged between 18 to 80 years old
* Patients presents with stable CAD or acute coronary syndrome (ACS)
* Eligible for percutaneous coronary intervention (PCI)
* Willing to provide DNA sample via blood drawn for genotyping and platelet reactivity assessment
* Willing and able to provide informed written consent

Exclusion Criteria:

* Primary PCI or rescue PCI
* Any urgent/emergent coronary angiography procedure that would not allow for genetic testing to be performed before PCI
* Failure of index PCI
* Patient or physician refusal to enroll in the study
* Patient with known CYP2C19 genotype prior to randomization
* Planned revascularization of any vessel within 30 days post-index procedure and/or of the target vessel(s) within 12 months post-procedure
* Anticipated discontinuation of clopidogrel or ticagrelor within the 12 months follow up period (e.g. for elective surgery)
* History of ischaemic or haemorrhagic stroke
* History of allergies to aspirin, ticagrelor, or clopidogrel
* Suffering from HIV or any blood transmitted disease.
* Considered at high risk of bleeding*
* Stage 5 chronic kidney disease (CKD) based on the National Kidney Foundation, Kidney disease quality outcome initiative (KDQOI) definition (Levey et al., 2005), or those who were on haemodialysis
* Pre-existing liver cirrhosis
* Pregnant women at any stage of gestation
* Patient is receiving immunosuppressive therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematous, etc.)
* Patient is receiving chronic anticoagulation therapy (i.e. vitamin K antagonist, direct thrombin inhibitor, Factor Xa inhibitor)
* Concomitant use of simvastatin/lovastatin >40 mg qd
* Concomitant use of potent CYP3A4 inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole) or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine)
* Non-cardiac condition limiting life expectancy to less than a year, per judgement of physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | From enrollment to 30 days post PCI
  Major adverse cardiovascular events (MACE) is defined as the composite of all-cause mortality, recurrent myocardial infarction (MI), repeat revascularization and stroke. The fourth universal definition of MI was used to retrospectively analyse recurrent MI. Any revascularization of the target coronary artery following the index incident, whether percutaneous or surgical, was referred to as repeat revascularization.

SECONDARY OUTCOMES:
Platelet Reactivity Index (PRI) | From enrollment to at least 2 weeks of maintenance dose
  Based on the PRI assessment, the participants can be categorised into treatment responders and non-responders. Clopidogrel and ticagrelor non-responses will be reported based on the cut-off point of PRI≥50%. For VASP method, a platelet reactivity index (PRI) of > 50% was defined as high on-treatment platelet reactivity (HTPR) which could lead to higher risk of ischaemic events post PCI, and a PRI of < 16% was defined as low on-treatment platelet reactivity (LTPR) which could lead to higher risk of bleeding. Hence, the optimal therapeutic window for antiplatelet therapy according to this VASP method is 17-49%

CONTACTS AND LOCATIONS:
Overall Officials: Nur Hafizah Annezah Utuh, Doctor of Philosophy (PhD), Principal Investigator — School of Pharmaceutical Sciences, Universiti Sains Malaysia
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided